CLINICAL TRIAL: NCT04138641
Title: Dutch Cangrelor Registry
Status: Completed | Type: Observational
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, A.H. Tavenier, R.S. Hermanides, Principal investigator, Isala
Other Study IDs: Dutch Cangelor registry
Record Dates: First submitted 2019-10-17; First posted 2019-10-24 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; NSTEMI - Non-ST Segment Elevation MI; Coronary Artery Disease
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Coronary Artery Disease | interventions — cangrelor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Cangrelor — Cangrelor intravenous

SUMMARY:
Cangrelor is a fast and directly acting platelet aggregation inhibitor. It is potentially indicated for several types of patients who are undergoing PCI. A nationwide cangrelor registry has up until now not been performed and with the introduction of cangrelor in the Netherlands its efficacy and safety will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* One of the following criteria:
* Patients naïve for P2Y12 inhibition undergoing PCI
* Patients with suboptimal P2Y12 inhibition undergoing PCI (patients who vomited after P2Y12 loading, out of hospital cardiac arrest (OHCA) patients with restoration of spontaneous circulation (ROSC), patients loaded with P2Y12 inhibitors though platelet inhibition still insufficient (<2 hours after oral loading dose)
* (N)STEMI patients loaded with P2Y12 inhibitors with large thrombus burden (thrombus grade 4 or 5) on initial coronary angiography (CAG) and undergoing primary PCI with expected insufficient P2Y12 inhibition

Exclusion Criteria:

* Patients on current/chronic treatment with P2Y12 inhibitors
* Patients (pre) treated with a GPI
* Patients with recent major bleeding complications or contraindication to dual antiplatelet therapy:
* hypersensitivity or allergy to and known contra-indication for aspirin, clopidogrel, ticagrelor or cangrelor
* history of major clinical bleeding or known coagulopathy
* active bleeding
* history of intracerebral mass, aneurysm, arteriovenous malformation, or hemorrhagic stroke
* known severe liver dysfunction
* Patients that received any organ transplant or are on a waiting list for any organ transplant
* Patients undergoing dialysis
* Pregnant or lactating female
* Patients currently participating in another investigational drug or device study

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing (primary) PCI
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
NACE | 48 hours
  The primary efficacy and safety endpoint is 48 hours Net Adverse Clinical Events (NACE), which is a composite endpoint of all-cause death (including cardiac death), recurrent myocardial infarction, target vessel revascularization, stroke, definite or probable stent thrombosis and bleeding (BARC type 2-5).

SECONDARY OUTCOMES:
NACE 30 days | 30 days
  Net Adverse Clinical Events (NACE), which is a composite endpoint of all-cause death (including cardiac death), recurrent myocardial infarction, target vessel revascularization, stroke, definite or probable stent thrombosis and bleeding (BARC type 2-5).
All individual endpoints in-hospital | In-hospital, mostly up to 72 hours.
  All individual endpoints in-hospital
All individual endpoints at 30-days | 30 days
  All individual endpoints at 30-days
TIMI 3 flow post PCI based on angiographic results | post-PCI, mostly up to 1 hour
  TIMI 3 flow post PCI

CONTACTS AND LOCATIONS:
Locations (1):
- R.S. Hermanides, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No